CLINICAL TRIAL: NCT06317571
Title: Evaluation of The Effect of Fertility Support Education Given to Infertile Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CelalBayarU-SBF-OT-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Infertility
Keywords: stress; cortisol Level; pregnancy Outcome; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Two groups with intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fertility support training (Experimental): The group will receive fertility support training.
  Interventions: Behavioral: fertility support education
- routine care (No Intervention): They will receive routine care.

INTERVENTIONS:
Behavioral: fertility support education — In the first module, female reproductive organs, the occurrence of pregnancy and the effect of stress on fertility are explained to women using models and training booklets. The effects of affirmation, which is one of the ways to positively affect the consciousness, and imagination, visualization and relaxation techniques, which are ways to positively affect the subconscious, on body and reproductive functions are explained. In the second module, women and their partners were also trained, and the effect of lifestyle on reproductive health was explained through the second module training booklet. In the third module, an example of a one-week program in which they could apply the methods described in the training before starting their treatments was introduced. In the fourth module, treatment process was explained to women and the practices described in the training were shared, which they could do to relax during this process.
  Arms: fertility support training

SUMMARY:
The aim of the this study was to evaluate the effect of fertility support education given to infertile couples before treatment.

DETAILED DESCRIPTION:
Before the treatment, couples were given fertility support training for four weeks. After the treatment was completed, the couples' stress level and quality of life, women's self-efficacy, fertility readiness, cortisol levels and pregnancy outcomes were examined.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with primary infertility
* have not received fertility support training before
* can speak Turkish

Exclusion Criteria:

* with psychiatric illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Infertility Stress Scale | two month
  This scale, which can be applied to both men and women, consists of three subscales and 14 items. The sub-dimensions of the scale are personal space, marital space and social space. A high score from the subscales of the scale indicates that stress has increased, while a low score indicates that stress has decreased.
Infertility Self-Efficacy Scale-Short Form | two month
  The scale was developed to evaluate the self-efficacy perceptions of infertile individuals about their cognitive, emotional and behavioral skill strengths. A 10-item short form of this scale, which consists of 16 items, was created in 2006. A minimum of 8 and a maximum of 32 points are obtained from the scale, and the higher the score obtained from the scale, the higher the perception of self-efficacy is considered.
Fertility Readiness Scale | two month
  The scale consists of three sub-dimensions: "Hope and Awareness", "Positive Emotions and Thoughts", and "Ready Body and Brain". Getting a high score on this scale indicates strong fertility readiness. The minimum score from the scale is 23 points and the maximum score is 115 points. The median score of this scale is 56 and it is stated that this score can be taken as the cut-off value. A score of 56 points or higher from the scale indicates that the woman feels more ready for pregnancy.
Fertiqol Quality of Life Scale | two month
  The scale evaluates quality of life. The core module consists of four dimensions: emotional, mind-body, relational and social, and the treatment module consists of two sub-dimensions: treatment environment and treatment tolerance. The total score of the scale varies between 0-100, and an increase in the total score indicates an increase in the quality of life.
Blood cortisol level | two month
  An increase in blood cortisol level indicates that stress increases, and a decrease indicates that stress decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Özge TOPSAKAL, PhD, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar Üniversitesi Hafsa Sultan Hastanesi, Manisa, Turkey (Türkiye)